CLINICAL TRIAL: NCT05027048
Title: Calcium Chloride for Prevention of Blood Loss From Uterine Atony During Intrapartum Cesarean Delivery (CALBLOC): a Double Blind, Randomized, Placebo Controlled Trial and Nested Population Pharmacokinetic and Pharmacodynamic Analysis
Brief Title: Calcium Chloride for Prevention of Blood Loss During Intrapartum Cesarean Delivery
Acronym: CALBLOC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other); Society for Obstetric Anesthesia and Perinatology (Other)
Responsible Party: Principal Investigator, Jessica Ansari, MD, MS, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 62206; MRTG-02-15-2022-Ansari (Other Grant/Funding Number: Foundation for Anesthesia Education and Research); YIG-2020 (Other Grant/Funding Number: Society Obstetric Anesthesia and Perinatology)
Record Dates: First submitted 2021-08-18; First posted 2021-08-30 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Uterine Atony; Uterine Atony With Hemorrhage; Postpartum Hemorrhage; Cesarean Section Complications
Keywords: calcium chloride; uterine atony; postpartum hemorrhage; cesarean delivery; intrapartum cesarean
MeSH Terms: conditions — Uterine Inertia; Postpartum Hemorrhage | interventions — Calcium Chloride

STUDY DESIGN:
Intervention Model Description: Double blind, placebo controlled randomized clinical trial with 1:1 allocation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, obstetrician, anesthesiologist, and clinical research staff will be blinded to the intervention. Drugs will be labeled only as "study drug"
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcium chloride (Experimental): 1 gram of calcium chloride in total volume 60mL with sterile saline, delivered over 10 minute controlled infusion at a constant rate (360mL/hour) beginning 2 minutes after fetal delivery and 1 minute after delayed cord clamp.
  This intervention occurs IN ADDITION TO standard care with oxytocin 2 unit bolus and infusion at 7.5 units per hour which begins immediately after fetal delivery.
  Interventions: Drug: Calcium chloride
- Saline placebo (Placebo Comparator): 60mL sterile saline, delivered over 10 minute controlled infusion at a constant rate (360mL/hour) beginning 2 minutes after fetal delivery and 1 minute after delayed cord clamp.
  This intervention occurs IN ADDITION TO standard care with oxytocin 2 unit bolus and infusion at 7.5 units per hour which begins immediately after fetal delivery.
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: Calcium chloride — See arm description above
  Arms: Calcium chloride
Drug: Saline placebo — see arm description above
  Arms: Saline placebo

SUMMARY:
Postpartum hemorrhage (PPH) is the leading cause of maternal morbidity and mortality worldwide. Up to 80% of PPH is caused by uterine atony, the failure of the uterine smooth muscle to contract and compress the uterine vasculature after delivery. Laboratory and epidemiological studies show that low extracellular and serum calcium levels, respectively, decrease uterine contractility. A pilot study performed by the investigators supports the hypothesis that intravenous calcium chloride is well tolerated and may have utility in preventing uterine atony. The proposed research will establish the relationship between uterine tone and calcium through a clinical trial with an incorporated pharmacokinetic and pharmacodynamic (PK/PD) study. In a randomized, placebo-controlled, double-blind trial, investigators will establish the effect of 1 gram of intravenous calcium chloride upon quantitative blood loss and uterine tone during cesarean delivery in parturients with high risk of uterine atony. Investigators will concurrently collect serial venous blood samples to measure calcium for PK/PD modeling in this pregnant study cohort. High-quality clinical research and development of novel therapeutics to manage uterine atony are critical to reduce the high maternal morbidity and mortality from PPH.

ELIGIBILITY:
Inclusion Criteria:

* Patient had a trial of labor for vaginal delivery prior to cesarean
* Patient received an oxytocin infusion for labor augmentation or induction prior to cesarean

Exclusion Criteria:

* renal dysfunction with serum Cr >1.0 mg/dL
* known underlying cardiac condition
* treatment with digoxin within the last 2 weeks for a maternal or fetal indication
* treatment with a calcium channel blocker medication within 24 hours
* hypertension necessitating intravenous antihypertensive medication within 24 hours
* emergent case in which study participation could in any way impede patient care by the judgement of the obstetrician, anesthesiologist, or bedside nurse

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ansari, MD, Principal Investigator — Stanford University
Locations (1):
- Jessica Ansari, Pacifica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole NM, Abushoshah I, Fields KG, Carusi DA, Robinson JN, Bateman BT, Farber MK. The interrater reliability and agreement of a 0 to 10 uterine tone score in cesarean delivery. Am J Obstet Gynecol MFM. 2021 May;3(3):100342. doi: 10.1016/j.ajogmf.2021.100342. Epub 2021 Feb 27. PMID 33652161
- [Result] Ansari JR, Yarmosh A, Michel G, Lyell D, Hedlin H, Cornfield DN, Carvalho B, Bateman BT. Intravenous Calcium to Decrease Blood Loss During Intrapartum Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2024 Jan 1;143(1):104-112. doi: 10.1097/AOG.0000000000005441. Epub 2023 Nov 3. PMID 37917943

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcium Chloride: 1 gram of calcium chloride in total volume 60mL with sterile saline, delivered over 10 minute controlled infusion at a constant rate (360mL/hour) beginning 2 minutes after fetal delivery and 1 minute after delayed cord clamp.
- Saline Placebo: 60mL sterile saline, delivered over 10 minute controlled infusion at a constant rate (360mL/hour) beginning 2 minutes after fetal delivery and 1 minute after delayed cord clamp.
Period: Overall Study
Arm/Group | Calcium Chloride | Saline Placebo
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Chloride | Saline Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (5.2) | 32.8 (5.2) | 33.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 24 | 19 | 43
  Hispanic or Latina | 17 | 23 | 40
  Non-hispanic black | 0 | 2 | 2
  Non-hispanic white | 16 | 12 | 28
  Other or declines to state | 3 | 4 | 7
Body Mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (4.6) | 32.2 (6.1) | 31.9 (5.4)
Gravida (n) [Median (Inter-Quartile Range); unit: pregnancies] — Number of prior pregnancies
  pregnancies | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
Para [Median (Inter-Quartile Range); unit: Prior pregnancies] — Number of prior pregnancies reaching 20 weeks and 0 days of gestation, regardless of the number of fetuses or the outcome
  Prior pregnancies | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1]
Gestational age (completed weeks) [Median (Inter-Quartile Range); unit: completed weeks] | 39 [39 to 40] | 39 [39 to 40] | 39 [39 to 40]
Advanced maternal age (n, %) [Count of Participants; unit: Participants] — Defined as age of >35 years at delivery
  Participants | 28 | 18 | 46
Hypertension from all causes (n, %) [Count of Participants; unit: Participants] | 7 | 17 | 24
Preeclampsia (n, %) [Count of Participants; unit: Participants] | 4 | 7 | 11
Diabetes, all causes (n, %) [Count of Participants; unit: Participants] | 7 | 11 | 18
Asthma (n, %) [Count of Participants; unit: Participants] | 3 | 7 | 10
Multiple gestation (n, %) [Count of Participants; unit: Participants] | 1 | 1 | 2
Chorioamnionitis (n, %) [Count of Participants; unit: Participants] | 9 | 8 | 17
Trial of Labor after Cesarean (TOLAC) (n, %) [Count of Participants; unit: Participants] | 5 | 3 | 8
Indication: first stage arrest [Count of Participants; unit: Participants] — Indication for cesarean delivery: failure of the first stage of labor (cervical dilation)
  Participants | 31 | 30 | 61
Indication: second stage arrest [Count of Participants; unit: Participants] — Indication for cesarean delivery: failure of the second stage of labor, also known as failure to descend. The cervical achieved full (10cm) dilation, but the fetus failed to descend with pushing to allow a vaginal delivery.
  Participants | 20 | 18 | 38
Indication: fetal intolerance of labor [Count of Participants; unit: Participants] — Indication for cesarean delivery: evidence of fetal distress with labor based upon analysis of the fetal heart tracing by the obstetrician.
  Participants | 16 | 18 | 34
Indication: failed operative vaginal delivery [Count of Participants; unit: Participants] | 1 | 3 | 4
Indication: maternal request [Count of Participants; unit: Participants] | 1 | 3 | 4
Indication: other [Count of Participants; unit: Participants] | 3 | 2 | 5
Maximum oxytocin dose in labor [Mean (Standard Deviation); unit: milliunits per minute] | 11.7 (8.5) | 12.4 (9.1) | 12.1 (8.8)
Hours of oxytocin exposure during labor [Mean (Standard Deviation); unit: hours] | 16.3 (12.0) | 18.5 (12.1) | 17.4 (12.1)

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Blood Loss
Description: Standardized volumetric and gravimetric assessment of blood loss during cesarean. Note: will analyze all participants, but planned subgroup analysis will also occur excluding patients with non-atonic reasons for blood loss including hysterotomy extension, placental abruption, cervical or vaginal laceration, etc
Time Frame: measurement occurs at conclusion of operating room case
Measure: Median (Inter-Quartile Range); unit: milliliters
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
milliliters | 840 [650 to 1434] | 1051 [796 to 1395]
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Test type: Superiority; p < 0.05, inverse Gaussian distribution and log li — a priori threshold for statistical significance p<0.05; Inverse Gaussian distribution and log link fit to estimate the effect size and 95% CIs; Mean Difference (Net) = 211, 95% CI 2-sided [-33 to 410] — Inverse gaussian regression with a log link was used to calculate the mean reduction in blood loss in the calcium group relative to placebo group

2. Secondary Outcome: Number of Participants With Postpartum Hemorrhage
Description: Postpartum hemorrhage was defined as quantitative blood loss > 1000 milliliters during operative course
Time Frame: operative course (within 4-6 hours of fetal delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
Participants | 24 | 34
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Test type: Superiority; Regression (poisson with robust SE); Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.48 to 1.03]

3. Secondary Outcome: Number of Participants With Second Line Uterotonic Requirement
Description: Yes/no: did the patient require treatment with methylergonovine, carboprost, and/or misoprostol for uterine atony
Time Frame: within 4 hours of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
Participants | 18 | 24
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Test type: Superiority; Poisson regression with robust SE; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.46 to 1.23]

4. Secondary Outcome: Number of Patients With a Transfusion Requirement
Description: Yes/no, if patient required transfusion of packed red blood cells prior to hospital discharge
Time Frame: 96 hours of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
Participants | 5 | 9
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Test type: Superiority; Risk Ratio (RR) = 0.56, 95% CI 2-sided [0.2 to 1.56]

5. Secondary Outcome: Change in Hematocrit From Baseline
Description: Measured pre-delivery hematocrit minus measured post-operative day 1 hematocrit. Correction factor of 3 hematocrit points per unit packed red blood cells transfused
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: Percentage of hematocrit
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
Percentage of hematocrit | 7.8 [6.6 to 9.2] | 9.6 [8.1 to 11.7]
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Test type: Superiority; Regression, Linear; Data were log transformed to approximate a normal distribution prior to linear regression; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-3.6 to 0.2]

6. Secondary Outcome: Total Oxytocin Bolus Requirement
Description: Total dose oxytocin bolus during cesarean
Time Frame: Cesarean duration, within 4-6 hours of fetal delivery
Population: Note: institutional standard policy is a 2 unit oxytocin bolus at the time of fetal delivery, with additional boluses prn
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
units | 3 [2 to 4] | 3 [2 to 4]

7. Secondary Outcome: Uterine Tone Numerical Rating Score, 7 Minutes After Fetal Delivery
Description: Uterine tone assessment: Obstetricians at the study institution use the following validated scale to grade uterine tone for all cesarean deliveries. The obstetrician places their hand directly on the uterine fundus and scores the adequacy of contraction. The interrater characteristics of this scale have been published (Cole et al, 2021).
  The scale ranges from 0-10. A score of 0 is the worst possible score and represents a flaccid, atonic uterus. A score of 10 is the best possible score and represents a firmly-contracted uterus.
Time Frame: 7 minutes after fetal delivery, 5 minutes after initiating study drug infusion
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
units on a scale | 7 [6 to 8] | 6.5 [6 to 7]
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Test type: Superiority; p = 0.415, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Uterine Tone Numerical Rating Score, 12 Minutes After Fetal Delivery
Description: Uterine tone assessment: Obstetricians at the study institution use the following validated scale to grade uterine tone for all cesarean deliveries. The obstetrician places their hand directly on the uterine fundus and scores the adequacy of contraction. The interrater characteristics of this scale have been published (Cole et al, PMID 33652161).
  The scale ranges from 0-10. A score of 0 is the worst possible score and represents a flaccid, atonic uterus. A score of 10 is the best possible score and represents a firmly-contracted uterus.
Time Frame: 12 minutes after fetal delivery, 10 minutes after initiating study drug infusion
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
units on a scale | 7 [6 to 8] | 7 [6 to 8]
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Test type: Superiority; p = 0.566, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Fluid Requirement
Description: Total crystalloid required during cesarean delivery in mL
Time Frame: Operating room duration, usually 2 hours
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
milliliters | 1594 (762) | 1502 (892)

10. Secondary Outcome: Percent Change in Mean Arterial Pressure
Description: Baseline mean arterial blood pressure recorded as average of first 6 mean arterial blood pressures recorded in operating room. Percent change calculated as measured mean arterial blood pressure minus baseline, divided by baseline. Reported here as the maximal decrease in mean arterial pressure. Repeated measures ANOVA reported in Statistical Analysis.
Time Frame: every 5 minutes for 30 minutes after study drug infusion initiation, compared to baseline
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
percent change | 16 [11 to 21] | 12 [4 to 20]
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Repeated measures ANOVA used to analyze differences between groups; Test type: Superiority; p = 0.348, ANOVA

11. Secondary Outcome: Percent Change in Heart Rate From Baseline
Description: Baseline heart rate recorded as average of first 6 heart rates recorded in operating room. Percent change calculated as measured heart rate minus baseline, divided by baseline. Maximal % increase in heart rate reported here. Repeated measures ANOVA used to analyze overall trend in Statistical Analysis below.
Time Frame: every 5 minutes for 30 minutes after study drug infusion initiation, compared to baseline
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
percent change | 0 [-4 to 5] | 10 [4 to 15]
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Repeated measures ANOVA used to assess for difference between groups in the % change from baseline heart rate; Test type: Superiority; p = 0.011, ANOVA; Repeated measures ANOVA

12. Secondary Outcome: Total Phenylephrine Requirement
Description: Total phenylephrine in milligrams administered while in the operating room
Time Frame: Duration of operating room time, up to 240 minutes
Population: Total of documented phenylephrine bolus and infusion administration during operative course
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 60 | 60
milligrams | 1.02 [0 to 2.26] | 1.09 [0.08 to 2.72]

13. Secondary Outcome: Pharmacokinetics of Calcium Chloride - Baseline Ionized Calcium
Description: Measured using an Abbott istat machine and CG8+ cartridge to determine venous blood gas ionized calcium levels
Time Frame: In the operating room prior to study drug administration (generally <30 minutes prior to fetal delivery and study drug administration)
Population: A total of 35 trial participants consented to provide serial blood specimens for ionized calcium measurement and pharmacokinetic analysis, per protocol.
Measure: Mean (Standard Deviation); unit: mmoL / liter
Groups:
- Calcium Chloride: 1 gram of calcium chloride in total volume 60mL with sterile saline, delivered over 10 minute controlled infusion at a constant rate (360mL/hour) beginning 2 minutes after fetal delivery and 1 minute after delayed cord clamp.
  This intervention occurs IN ADDITION TO standard care with oxytocin 2 unit bolus and infusion at 7.5 units per hour which begins immediately after fetal delivery.
  Calcium chloride: See arm description above
- Saline Placebo: 60mL sterile saline, delivered over 10 minute controlled infusion at a constant rate (360mL/hour) beginning 2 minutes after fetal delivery and 1 minute after delayed cord clamp.
  This intervention occurs IN ADDITION TO standard care with oxytocin 2 unit bolus and infusion at 7.5 units per hour which begins immediately after fetal delivery.
  Saline placebo: see arm description above
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 19 | 16
mmoL / liter | 1.15 (0.02) | 1.16 (0.03)
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Test type: Superiority; p = 0.25, t-test, 2 sided

14. Secondary Outcome: Pharmacokinetics of Calcium Chloride - Peak Change in Ionized Calcium From 1 Gram of Calcium Chloride
Description: Generated from a 2-compartment population pharmacokinetic model in NONMEM using serial venous blood gas ionized calcium concentrations.
Time Frame: At Tmax (conclusion of the 10-minute intravenous calcium chloride infusion
Population: Participants who participated in the nested pharmacokinetic study and were randomly assigned to the calcium chloride group.
Measure: Mean (95% Confidence Interval); unit: mmoL / liter
Groups:
- Pharmacokinetic Subgroup: Calcium Chloride Recipients: Subgroup of participants who agreed to venous blood sampling for ionized calcium measurement for pharmacokinetic analysis and were assigned to receive calcium chloride (not placebo)
Arm/Group | Pharmacokinetic Subgroup: Calcium Chloride Recipients
Number analyzed (Participants) | 18
mmoL / liter | 0.39 [0.37 to 0.42]
Statistical Analysis 1: Comparison: Pharmacokinetic Subgroup: Calcium Chloride Recipients; Test type: Other; Note: a two-compartment pharmacokinetic model was generated in NONMEM using 6 venous blood ionized calcium measurements per participant at random times. The change in ionized calcium was defined as a measured value minus the measured baseline for the patient. Once the two-compartment pharmacokinetic model was generated, NONMEM was used to generate a predicted ionized calcium concentration at 10 minutes (Tmax) for each participant to generate mean and 95% confidence interval

15. Secondary Outcome: Pharmacodynamic Effect of Calcium Upon Uterine Tone NRS
Description: Data were not collected. This measure required blood specimens to be obtained at the time of tone scores and this was not done.
Time Frame: Within 20 minutes of study drug administration
Population: Data not collected (unable to obtain blood specimens at the time of tone scores)
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Quantitative Blood Loss, Subgroup Quantitative Blood Loss (QBL, mL), Excluding Cases of Documented Non-atonic Bleeding
Description: Pre-specified subgroup analysis of primary outcome:
  Because the proposed mechanism of calcium action-improving uterine contractility-was not expected to improve bleeding from causes such as hysterotomy extension or arterial bleeding, the trial was powered for a prespecified subgroup analysis excluding patients with nonatonic blood loss documented in the surgeon's operative report. Documented nonatonic bleeding was defined as presence in the surgeon's operative report narrative of any of the following: hysterotomy extension, hysterotomy types other than low transverse (eg classical, T- or J-shaped), invasive or abnormally adherent placenta, placental abruption, uterine rupture, bleeding from leiomyomas, grade 3 or 4 vaginal lacerations, or cervical lacerations.
Time Frame: Calculated at conclusion of operating room case
Population: Pre=specified subgroup analysis, excluded cases of documented nonatonic bleeding (mostly due to hysterotomy extension, present in 21 participants allocated to calcium and 20 participants allocated to placebo).
Measure: Median (Inter-Quartile Range); unit: milliliters
Arm/Group | Calcium Chloride | Saline Placebo
Number analyzed (Participants) | 39 | 40
milliliters | 759 [592 to 912] | 922 [754 to 1193]
Statistical Analysis 1: Comparison: Calcium Chloride vs Saline Placebo; Test type: Superiority; p < 0.05, Inverse Gaussian regression, log link; Mean Difference (Net) = 356, 95% CI 2-sided [159 to 515] — Reduction in blood loss was calculated by inverse Gaussian regression with a log link as detailed in the description of statistical methods for the primary outcome

ADVERSE EVENTS:
Time Frame: Day of cesarean delivery (and study drug administration). Adverse events were assessed formally at the conclusion of the operating room course prior to transport to the recovery unit. The clinical anesthesiologist discussed all possible side effects with the patient prior to filling out a form. (Anesthesiologist and patient blinded to allocation).
Arm/Group | Calcium Chloride | Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 23/60 | 25/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcium Chloride (N=60) | Saline Placebo (N=60)
New or subjective worsening in nausea (Gastrointestinal disorders) | 18 (18) | 18 (18)
New or increased vomiting (Gastrointestinal disorders) | 12 (12) | 11 (11) — If patient began vomiting or experienced subjective worsening after initiating study drug infusion.
Intravenous line pain (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Burning or discomfort at or proximal to the site of the intravenous line
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) — Patient perception of hot or flushed skin
Change in heart rate (Cardiac disorders) | 1 (1) | 6 (6) — Clinically significant changes in heart rate for which the anesthesiologist administered a treatment medication (ie glycopyrrolate, epinephrine, or atropine for bradycardia, beta blockade, phenylephrine, etc for tachycardia)
Severe range hypertension (Cardiac disorders) | 0 (0) | 1 (1) — Hypertension (>160mmHg systolic or >100mmHg diastolic) resulting in treatment with an intravenous antihypertensive agent
Abnormal tastes or sensations (Nervous system disorders) | 0 (0) | 2 (2) — Patient note of any abnormal tastes or subjective abnormal sensations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT05027048/Prot_SAP_000.pdf